CLINICAL TRIAL: NCT01607619
Title: A 12-week Multi-site Trial of the Dietary Supplement Anatabine (RCP006) to Determine the Effects on Peripheral Markers of Inflammation in Patients With Elevated Levels of C-reactive Protein (CRP)
Brief Title: Effect of Anatabine on Elevated Blood Levels of C-reactive Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roskamp Institute Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: RI-11-01
Record Dates: First submitted 2012-02-03; First posted 2012-05-30 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Inflammation
Keywords: CRP
MeSH Terms: conditions — Inflammation | interventions — anatabine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: Anatabine — 1mg anatabine in a mint-flavored mannitol lozenge
  Other Names: RCP006

SUMMARY:
The investigators are studying a dietary supplement called anatabine in a lozenge form named RCP006. The main purpose of this study is to evaluate the effects of this dietary supplement on normal human inflammatory function. The investigators will see this effect in volunteers who have markers of higher levels of inflammation to begin with. The investigators anticipate that anatabine will reduce markers of inflammation. Therefore the investigators are looking for volunteers with high blood levels of C-reactive Protein (CRP) and will monitor the blood CRP levels at several time points throughout the study.

DETAILED DESCRIPTION:
The investigators are studying a dietary supplement called anatabine which for the purposes of this study has been made into lozenges and named RCP006. Anatabine, the only active ingredient of RCP006, occurs throughout the world in the human food chain. Anatabine has been in the human food supply and in human use for centuries. Humans are exposed to anatabine in tobacco products and common and widely consumed food crops such as potatoes, peppers, eggplants and tomatoes. The main purpose of this study is to evaluate the effects of this dietary supplement on normal human inflammatory function. Compounds that are chemically similar to anatabine have been shown to reduce inflammatory responses, and laboratory studies show anti-inflammatory properties for anatabine. The investigators want to explore this further in human studies to see if anatabine can maintain normal levels of inflammatory function. The investigators will see this effect more easily if the investigators look at the effects of anatabine in volunteers who have markers of higher levels of inflammation to begin with. The investigators anticipate that anatabine will reduce markers of inflammation. To look for inflammation the investigators will test blood levels of a protein called C-reactive protein. C-reactive protein (CRP) is a protein found in the blood, the levels of which rise in response to inflammation. Therefore the investigators are looking for volunteers with high blood levels of CRP and will monitor the blood CRP levels at several timepoints throughout the study. The investigators will also collect blood samples to measure other indicators of inflammation, and to measure blood levels of anatabine.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults with elevated blood levels of hsCRP

Exclusion Criteria:

* pregnancy or planning pregnancy
* current tobacco use
* current steroid use
* allergy to study product components

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Blood levels of hsCRP | Days 1, 14, 42, 70

SECONDARY OUTCOMES:
Blood levels of inflammatory markers | Days 1, 14, 42, 70

CONTACTS AND LOCATIONS:
Overall Officials: Dale Wilson, MD, Principal Investigator — McLaren Community Medical Center; Vittorio Morreale, MD, Principal Investigator — Medical Practice, Shelby Township
Locations (3):
- United States (3):
  - The Roskamp Institute, Inc., Sarasota, Florida
  - McLaren Community Medical Center, Flint, Michigan
  - Medical Practice, Shelby, Michigan